CLINICAL TRIAL: NCT02396485
Title: Early Versus Late Feeding After Cesarean Delivery: A Randomized Controlled Trial
Brief Title: Early Feeding After A Cesarean Delivery Hastens Recovery Time for Bowel Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 13-0391
Record Dates: First submitted 2015-02-26; First posted 2015-03-24 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Gastrointestinal Disorders, Functional
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early Feeding Arm (Experimental): Patients will be started on regular diet within 6 hrs postoperative.
  Interventions: Other: Regular diet within 6hrs postoperative
- Late Feeding Group (No Intervention): Patients will be remaining nothing per os (NPO, i.e nothing per mouth) for 12hrs, and the diet then advanced as tolerated after 12hrs as standard postoperative protocol in the investigators' institution.

INTERVENTIONS:
Other: Regular diet within 6hrs postoperative — Patients will be randomized to regular diet within 6 hrs postoperative (Early group) versus remaining nothing per os (NPO, i.e nothing per mouth) for 12hrs, and the diet then advanced as tolerated after 12hrs (Routine Group) as standard postoperative protocol in the investigators' institution.
  Arms: Early Feeding Arm

SUMMARY:
After institutional review approval, pregnant women that are scheduled for elective cesarean delivery will be approached for participation in the study. The study informed consent will be obtained. The study's time frame inclusive will be from 2013 till 2016.

Patients will be randomized to regular diet within 6 hrs postoperative (Early group) versus remaining nothing per os (NPO, i.e nothing per mouth) for 12hrs, and the diet then advanced as tolerated after 12hrs (Routine Group) as standard postoperative protocol in the investigators' institution.

Primary outcome will be time to pass flatus. Secondary outcomes will include hospital length of stay, postoperative nausea, vomiting and patient satisfaction. Randomization will be performed using a computer generated random list of numbers assigning patients to the 2 groups of the study. This list of random number assignments will be kept secure in an opaque envelope until the end of the study. Patients in the Early group will be started on regular diet within 6 hrs of surgery, whereas the routine group patients will be kept strict NPO 12hrs, and clear liquid diet will be started after 12hrs. Diet will be advanced as tolerated, i.e. if clears were tolerated or flatus or bowel movement occurred, patients will be started on solid foods. If diet not tolerated, a full liquid diet will be given instead. Consequently if patient tolerated full liquid diet, a regular diet will be then initiated. Patients will be discharged home only if they tolerate solid food with absence of emesis, have flatus or bowel movement. Time Zero is defined as time of skin incision.

DETAILED DESCRIPTION:
After institutional review approval, pregnant women that are scheduled for elective cesarean delivery will be approached by Principal investigator or any of the co-investigators for participation in the study during the the preoperative visit which coincides with the same day of scheduled cesarean in a private patient room. . Prospective subjects will be presenting for their preoperative appointment (same day of scheduled cesarean delivery) in labor and delivery and will be asked to participate in the study. The study will be explained as in the consent form and if agreed patients will elect either to or not to participate in the study after all risks and benefits are explained. Data to be collected will consist of time in minutes of passing flatus, time in minutes of having a bowel movement, hospital length of stay, postoperative nausea, vomiting and presence of ileus (unable to tolerate diet, abdominal distention, no bowel movement nor flatus, abdominal x-ray demonstrating air/fluid levels in bowel). Patients will be contacted once to twice a day for assessment of data points mentioned above. If elected to participate consents will be obtained. Randomization will be done at time of consents. The study's time frame inclusive will be from 2013 till 2016.

ELIGIBILITY:
Inclusion Criteria:

* Gravid women greater than 37 weeks undergoing elective cesarean delivery.

Exclusion Criteria:

* Intra-operative bowel surgery
* Preeclampsia requiring magnesium sulfate
* Diabetes Mellitus.
* Planned secondary closure of the skin incision
* Any gastrointestinal and/or medical conditions that precludes early consumption of solid food
* General anesthesia
* Gestational age less than 37 weeks.
* Patients who are mentally incapacitated or decisionally impaired.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 177 (Actual)
Dates: Start 2014-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Passing Flatus | participants will be followed for the duration of hospital stay, an expected average of 2-5 days
  The primary outcome is the duration in minutes from surgery completion(skin closure) and time of passage of first flatus (passing gas per anus).

SECONDARY OUTCOMES:
Bowel sounds | participants will be followed for the duration of hospital stay, an expected average of 2-5 days
  First time in minutes from completion of surgery that bowel sounds are heard active.
Bowel Evacuation | participants will be followed for the duration of hospital stay, an expected average of 2-5 days
  First time in minutes from completion of surgery that patient reports passing bowel movement or stools.
Nausea or vomiting | participants will be followed for the duration of hospital stay, an expected average of 2-5 days
  First time in minutes from completion of surgery that patient reports nauseated or has actually had emesis.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio F Saad, MD, Principal Investigator — UTMB Galveston Texas

REFERENCES:
- [Background] Hsu YY, Hung HY, Chang SC, Chang YJ. Early oral intake and gastrointestinal function after cesarean delivery: a systematic review and meta-analysis. Obstet Gynecol. 2013 Jun;121(6):1327-1334. doi: 10.1097/AOG.0b013e318293698c. PMID 23812470
- [Background] Bar G, Sheiner E, Lezerovizt A, Lazer T, Hallak M. Early maternal feeding following caesarean delivery: a prospective randomised study. Acta Obstet Gynecol Scand. 2008;87(1):68-71. doi: 10.1080/00016340701778849. PMID 18158630
- [Background] Patolia DS, Hilliard RL, Toy EC, Baker B. Early feeding after cesarean: randomized trial. Obstet Gynecol. 2001 Jul;98(1):113-6. doi: 10.1016/s0029-7844(01)01387-4. PMID 11430967
- [Derived] Saad AF, Saoud F, Diken ZM, Hegde S, Kuhlmann MJ, Wen TS, Hankins GD, Saade GR, Costantine MM. Early versus Late Feeding after Cesarean Delivery: A Randomized Controlled Trial. Am J Perinatol. 2016 Mar;33(4):415-9. doi: 10.1055/s-0035-1565918. Epub 2015 Oct 19. PMID 26479169